CLINICAL TRIAL: NCT04042454
Title: A Randomized, Controlled Study to Evaluate the Safety and Tolerance of an Infant Formula With Locust Bean Gum in Infants With Regurgitation
Brief Title: To Assess the Safety and Tolerance of Infant Formula With Locust Bean Gum in Infants With Regurgitation
Acronym: Solar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBB18TA19425
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2021-09

CONDITIONS: Regurgitation, Gastric; Diarrhea
MeSH Terms: conditions — Laryngopharyngeal Reflux; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (Experimental): Cow's milk-based infant formula containing the thickener locust bean gum containing prebiotic oligosaccharides and postbiotics
  Interventions: Other: milk based anti-regurgitation infant formula
- Control Product (Active Comparator): Cow's milk-based infant formula containing prebiotic oligosaccharides and postbiotics
  Interventions: Other: Milk based infant formula

INTERVENTIONS:
Other: milk based anti-regurgitation infant formula — Cow's milk-based infant formula containing the thickener locust bean gum containing prebiotic oligosaccharides and postbiotics for a period of 8-14 weeks (dependent on infants age at baseline). The intervention last's until the infant's age of 17 weeks.
  Arms: Test Product
Other: Milk based infant formula — Cow's milk-based infant formula containing prebiotic oligosaccharides and postbiotics for a period of 8-14 weeks (dependent on infants age at baseline). The intervention last's until the infant's age of 17 weeks.
  Arms: Control Product

SUMMARY:
A randomized, controlled study to evaluate the safety and tolerance of an infant formula with locust bean gum in infants with regurgitation. (Solar)

ELIGIBILITY:
Inclusion Criteria:

1. Singleton infants with regurgitation who are otherwise healthy
2. Diagnosed with regurgitation according to the (adapted) Rome IV diagnostic criteria.
3. Term infants with a gestational age at birth of ≥37 weeks + 0 days and ≤41 weeks + 6 days
4. Aged > 3 weeks (21 days) and < 9 weeks (63 days) at screening
5. Exclusively formula fed for ≥ 7 days before screening
6. Written informed consent from the parent(s) and/or legally acceptable representative(s)

Exclusion Criteria:

1. Low birth weight for gestational age and gender
2. Infants diagnosed with or suspected to have gastroesophageal reflux disease (GERD). I
3. Infants who received any of the following medication within 4 weeks prior to screening: systemic antibiotics, prokinetics and/or proton pump inhibitors and/or (other) medication to treat regurgitation
4. Infants who already consumed a thickened anti-regurgitation (AR) formula or used thickening supplements
5. Infants who already started complementary feeding
6. Infants with a gastrointestinal infection within 4 weeks prior to screening
7. Infants with a congenital condition, previous or current illness, and/or medication use that could interfere with the main study outcomes according to the investigator
8. Infants known or suspected to have: allergy for fish, soy protein, soy oil or corn; lactose intolerance; galactosaemia including history of any other allergic manifestations or known allergy to any of the study product ingredients and/or requiring a fibre-free diet
9. Infants known or suspected to have allergy to cow's milk protein
10. Presence of any other gastrointestinal symptom(s)/disorder(s) that are not functional in nature, as assessed by the investigator's clinical judgement
11. Participation in any other studies involving investigational or marketed products concomitantly or prior to screening
12. Incapability of the parent(s) to comply with the study protocol or investigator's uncertainty about the willingness or ability of the parent(s) to comply with the protocol requirements

Ages: 3 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Average stool consistency | 8 weeks
  The average stool consistency (based on the 4-point Brussels Infant and Toddler Stool Scale [BITSS]) of the 8th week of intervention, adjusted for the baseline stool consistency score. Catagories are hard stools, formed stools, loose stools and watery stools. https://bitss-stoolscale.com/ (assessed 31-Jan-19) can be used as a further reference.

SECONDARY OUTCOMES:
To assess the average stool consistency | 8 weeks
  The average stool consistency based on the BITSS, adjusted for baseline, for every week until the 8th week of intervention and for the week prior to the age of 17 weeks
The average stool frequency | 8 weeks
  The average stool frequency, adjusted for baseline, for every week until and including the 8th week of intervention and for the week prior to the age of 17 weeks
Incidence of diarrhoea: | 8 weeks, 17 weeks
  1. based on the WHO criteria and derived from the BITSS, for every week (until and including week 8 of intervention, and at the age of 17 weeks)
  2. based on investigator's diagnosis of diarrhoea (throughout the entire study)
IGSQ sum and individual item scores | 2, 4, 8, 17 weeks
  IGSQ sum and individual item scores, adjusted for baseline, at 2, 4 and 8 weeks of intervention, and at the age of 17 weeks
Gut microbiota composition and function | 17 weeks
  Gut microbiota composition and function (acetate, lactate, pH, calprotectin, ammonium and sIgA) at baseline and at the age of 17 weeks
Regurgitation | 2,4,8,17 weeks
  Regurgitation: number of regurgitation episodes per day and the regurgitation volume score, adjusted for baseline, at 2, 4 and 8 weeks of intervention, and at the age of 17 weeks (based on 3-day diaries)

CONTACTS AND LOCATIONS:
Locations (16):
- Italy (5):
  - A.O.U. Ospedali Riuniti di Ancona, Ancona
  - Ospedale pediatrico Giovanni XXIII, Bari
  - Azienda Ospedaliera Universitaria G. Martino, Messina
  - Ospedale dei bambini Buzzi, Milan
  - Ospedale F. Del Ponte, Varese
- Poland (6):
  - Poliklinika Ginekologiczno-Położnicza Sp. z o.o. Sp. k., Bialystok
  - Osrodek badan Klinicznych IN-VIVO sp. z o.o., Bydgoszcz
  - Gabinet Lekarski, Rzeszów
  - NZLA Michalkowice Jarosz, Siemianowice Śląskie
  - Alergo-Med Specjalistyczna Przychodnia Lekarska sp. z o.o, Tarnów
  - EPOKA Niepubliczny Zaklad Opieki Zdrowotnej Piotr Chodkiewicz Sp. z o.o, Żnin
- Ukraine (5):
  - Communal Nonprofit Enterprise "City Children's Clinical Hospital, Dnipro
  - Communal Nonprofit Enterprise "City Children's Clinical Hospital, Kharkiv
  - Communal Nonprofit Enterprise "Lviv City Children's Clinical Hospital", Lviv
  - Communal Enterprise "Poltava Regional Children's Clinical Hospital of Poltava Regional Council, Poltava
  - Communal Non-Profit Enterprise of Sumy Regional Council "Regional Children Clinical Hospita, Sumy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] ESPGHAN 55th Annual Meeting Abstracts. J Pediatr Gastroenterol Nutr. 2023 Jun 1;76(S1 Suppl 1):1-1407. doi: 10.1097/MPG.0000000000003823. Epub 2023 May 19. No abstract available. PMID 37204764